CLINICAL TRIAL: NCT04980131
Title: Application of 3-Dimensional Printing Guide Template and Pointed Lotus-style Regulator in Percutaneous Pedicle Screw Fixation for Thoracolumbar Fractures
Brief Title: Application of 3-Dimensional Printing Guide Template and Pointed Lotus-style Regulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ming Zhang (Other)
Collaborators: The Second People's Hospital of Huai'an (Other)
Responsible Party: Sponsor-Investigator, Ming Zhang, medium-grade professional title, The Second People's Hospital of Huai'an
Organization: The Second People's Hospital of Huai'an (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HEYLL201705
Record Dates: First submitted 2021-07-08; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Vertebral Fracture
Keywords: 3D printing guide template; pointed lotus-style regulator; thoracolumbar compression fracture; percutaneous pedicle screw fixation
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Experimental): Group C were received PPSF with pointed lotus-style regulator
  Interventions: Device: Pointed lotus root regulator and guide template aided PPSF
- Group B (Experimental): Group B were received PPSF with Flat ended lotus root regulator
  Interventions: Device: Flat ended lotus root regulator and guide template aided PPSF
- Group A (No Intervention): Group A were received traditional PPSF

INTERVENTIONS:
Device: Pointed lotus root regulator and guide template aided PPSF — 20 patients in group C received PPSF with pointed lotus-style regulator
  Arms: Group C
Device: Flat ended lotus root regulator and guide template aided PPSF — 20 patients in group B received PPSF with flat ended lotus-style regulator
  Arms: Group B

SUMMARY:
This study aims to analysis the efficacy of the 3D printing percutaneous guide template in combination with the pointed lotus-style regulator in percutaneous pedicle screw fixation.

DETAILED DESCRIPTION:
All thoracolumbar fractures patients receiving percutaneous pedicle screw fixation (PPSF) were enrolled and randomly divided into 3 groups. Patients in Group A received traditional PPSF, while patients in Group B received PPSF with flat end lotus-style regulator and patients in Group C received PPSF with pointed lotus-style regulator.

ELIGIBILITY:
Inclusion Criteria:

* The thoracolumbar vertebral compression fracture which the injury time is less than 7 days
* The vertebral fracture sites where are located in T11-L2
* No clinical neurological symptoms and signs
* The patients who have complete preoperative X-ray, CT, MRI and other imaging data

Exclusion Criteria:

* Vertebral burst fracture with spinal canal occupation
* Fracture caused by severe osteoporosis or tumor and other pathological factors
* Moderate and severe scoliosis
* Patients with pedicle dysplasia
* Patients with severe heart, liver and kidney diseases, diabetes, immune diseases, mental diseases who cannot tolerate surgery
* Coagulation dysfunction or surgical site of the skin infection

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
First puncture success rate,number of insertions before reaching the desired position, number of fluoroscopy before reaching the desired position, radiation dosage before reaching the desired position, operation time before reaching the desired position | twenty months
  All the operations were successfully completed. The number of pedicles successfully first pierced in group C was higher than that in group A and group B (P<0.05);The number of insertion, fluoroscopy and operation time before the insertion needle reached the ideal position, the total number and time of intraoperative fluoroscopy, and the intraoperative blood loss in group C were all significantly lower than those of group A and group B (P<0.05)
VAS scores after surgery | twenty-two months
  All patients were followed up 6 months after surgery. VAS scores at 1 day and 7 days after surgery were higher in Group A than those in other groups（P<0.05）, but no differences were found VAS scores at 1 , 3 and 6 months after surgery in 3 groups.Specific methods: drawing a 10cm line on the paper, one end of the horizontal line is 0, that is painless; The other end is 10, which means severe pain; The intermediate part indicates different levels of pain. Asking the patient to mark the level of pain on a horizontal line according to how he or she feels. 0-2: meaning comfortable; 3-4: slight discomfort; 5-6: moderate discomfort; 7-8: Severe discomfort;9-10: Extreme discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Quan Zhou, Zhou, Study Director — The Second People's Hospital of Huai'an
Locations (1):
- The Huai'an Second People's Hospital, Huai'an, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Wait for the results of related parallel trials before considering sharing data

REFERENCES:
- [Result] Zhang M, Li J, Fang T, Zhao J, Pan W, Wang X, Xu J, Zhou Q. Evaluation of a Three-Dimensional Printed Guide and a Polyoxymethylene Thermoplastic Regulator for Percutaneous Pedicle Screw Fixation in Patients with Thoracolumbar Fracture. Med Sci Monit. 2020 Jan 14;26:e920578. doi: 10.12659/MSM.920578. PMID 31932574
- [Derived] Zhang M, Li J, Fang T, Yan J, Wu L, Zhou Q. Application of 3-dimensional printing guide template and pointed lotus-style regulator in percutaneous pedicle screw fixation for thoracolumbar fractures. Sci Rep. 2022 Feb 21;12(1):2930. doi: 10.1038/s41598-022-06256-x. PMID 35190566
- See also: This work is licensed under Creative Common AttributionNonCommercial-NoDerivatives 4.0 International (CC BY-NC-ND 4.0) — http://www.medscimonit.com/abstract/index/idArt/920578

DOCUMENTS (1):
  • Informed Consent Form (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT04980131/ICF_000.pdf